CLINICAL TRIAL: NCT02476396
Title: Structural Stability of Carotid Plaque and Symptomatology
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0289; A535700 (Other: UW Madison); SMPH\NEURO SURG\NEURO SURG (Other: UW Madison); 1F31HL141008-01A1 (NIH); 1R01HL147866-01A1 (NIH); R01NS064034 (NIH); Protocol Version Aug 2023 (Other: UW Madison)
Record Dates: First submitted 2015-06-05; First posted 2015-06-19 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Carotid Stenosis; Stroke; Carotid Artery Plaque; Transient Ischemic Attack; Cerebrovascular Accident; Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis; Stroke; Ischemic Attack, Transient | interventions — Endarterectomy, Carotid; Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects and controls will have 2 tubes of blood drawn. DNA will be removed and may be saved for future testing. Some cells from the participant's blood may be kept alive and growing in the laboratory as a "cell line". Creating a cell line will allow the investigators to get more DNA for future research.
  Subjects will have their carotid plaques removed via standard carotid endarterectomy. This surgical procedure is part of the standard clinical care.
  Blood samples will be decoded and unidentifiable, kept in a secure freezer box (with a lock and key) and stored in chamber of 1 -800C freezer used only to store human blood and RNA samples.
  Plaque specimens will be de-identified. Samples will be kept in a secure freezer box stored in a chamber with authorized access only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient-subject: Patients will be recruited from the population of patients scheduled to undergo carotid endarterectomy or stenting (endovascular) for established clinical indications. These indications include patients scheduled to have a carotid endarterectomy or stenting due to the presence of a high-grade atherosclerotic cervical internal carotid artery stenosis with or without clinical symptoms, following the ACAS or NASCET criteria (carotid artery stenosis of 60% or greater without clinical symptoms; stenosis 70% or greater with clinical symptoms).
  Interventions: Procedure: Carotid Endarterectomy or Stenting
- patient-control: The controls will be recruited by the patient-subjects. The investigators will ask their patient-subjects to speak to a spouse or family member to see if they are interested in participating. If they do have an interest they will contact the research team/study coordinator(s). In case, a spouse or a family member is accompanying the patient-subject, they will be recruited at the same time as the patient-subject.

INTERVENTIONS:
Procedure: Carotid Endarterectomy or Stenting — Carotid endarterectomy is a procedure to treat carotid artery disease. This disease occurs when fatty, waxy deposits build up in one of the carotid arteries. The carotid arteries are blood vessels located on each side of your neck (carotid arteries).
  This buildup of plaques (atherosclerosis) may restrict blood flow to your brain. Removing plaques causing the narrowing in the artery can improve blood flow in your carotid artery and reduce your risk of stroke.
  In carotid endarterectomy, you an anesthetic. Your surgeon makes an incision along the front of your neck, opens your carotid artery and removes the plaques that are clogging your artery. Your surgeon then repairs the artery with stitches or a patch made with a vein or artificial material (patch graft).
  Source: Mayo Clinic
  Carotid stenting uses a expandable metal coil to prevent the artery from narrowing.
  Groups: patient-subject

SUMMARY:
The purpose of the research is to understand structural plaque abnormalities that make a carotid plaque unstable and brake off (embolize) which would help to predict and treat individuals who are likely to suffer not only classic episodic major strokes but also cognitive impairment.

DETAILED DESCRIPTION:
This study examines the relationship between the structural stability of carotid atherosclerotic plaque forming at the bifurcation of the common internal/external carotids and the ability of such lesions to cause disease. The theory behind this work is the hypothesis that carotid atherosclerotic stroke presents not only as a classical episodic clinical condition, but may also involve elements of a continuous process involving large and small vessel circulations, microcirculatory changes, cellular metabolic resistance to ischemia and micro embolic events. Recent studies suggest for every recognized clinical stroke, 5 silent strokes take place.

The patient implications are enormous as imaging suggests 11 million "silent strokes" occur yearly in the US with poor understanding of the pathophysiology or cognitive consequences for our patients. Within this framework, the investigators choose to study the hypothesis that carotid artery atherosclerosis is likely to cause microemboli, as well as classic macroemboli, which may result in more subtle disturbances than those ordinarily detected by more obvious clinical events such as stroke and transient ischemia attacks.

Understanding the structural plaque abnormalities that render a carotid plaque unstable and at risk of embolization would help to predict and treat individuals who are likely to suffer not only classic episodic major strokes, but also cognitive impairment from the contribution of microemboli to this overall disease process. The investigators have previously described a non-invasive ultrasound-based measure of plaque structural stability which will be further studied in this proposal. This study will expand on previous work performed at the University of Wisconsin-Madison, and will include patients with carotid artery stenosis, both with and without classic stroke symptoms, as well as a control group of patients without known atherosclerotic disease. Current treatments for carotid artery stenosis include either carotid endarterectomy to remove plaque or carotid stenting using a expandable metal coil to prevent the artery from narrowing.

In the previous version of this protocol, the investigators have enrolled 95 -subjects (75 patient-subjects and 20 control-subjects) with no safety concerns. Findings include new understanding of the relatively of atherosclerosis and cognition as well as the basic pathophysiology of atherosclerotic large to small vessel disease.

The study will run for 5 years from IRB approval with potential to further expand it. All patient-subjects will have a baseline and 1-year follow-up, ultrasound, TCD, blood collection and cognitive study to see if endarterectomy or stenting (endovascular) affected pre-op change. Change in cognition will be compared to report studies in the normal control group. In past, carotid patients have been recruited at a greater pace. Given the complexity of these studies the investigators anticipate recruitment and complete analysis of 20 patients/year. During this time initial psychological testing will be done pre-operatively. During the final year of the study, the data analysis of the plaque ultrasounds, and histopathology and 1-year follow-up the patient received in the last year of recruitment will take place. The investigators can recruit additional patients to fill any missing data points if these results identify a subset of classically asymptomatic patients with significant carotid plaques and microemboli causing vascular cognitive decline.

* Specific Aim 1: Atherosclerosis, plaque elasticity, strain defects and histopathology of plaque. This aim will study the relationship of structural instability in the carotid plaques with histopathologic evidence for fissuring of the plaques that may represent a micro-emboli source. The determination of a structural defect causing abnormal strain measurements in a carotid atherosclerotic plaque will be important in understanding the pathophysiology of this disorder, as well as, addressing future treatment strategies, which could include preventing angiogenesis, thrombosis, or abnormal cholesterol deposit within the plaque.
* Specific Aim 2: Plaque strain deficits and microemboli. In this aim, the investigators will preoperatively measure the structural stability of each plaque ultrasonically while simultaneously recording distally for the presence of microemboli over time within the carotid system. Statistical analysis will establish the structural instability signature that predicts ongoing subclinical microemboli.
* Specific Aim 3: Plaque strain deficits, microemboli, and cognition. This aim will analyze increased elasticity strain within carotid plaques as measured preoperatively with ultrasound and correlate these parameters with cognition
* Specific Aim 4: Blood RNA expression profiles can be used as biomarkers to identify the patients with a higher risk of plaque instability. This aim will analyze the mRNA and microRNA expression profiles of the blood and the excised plaque samples from patients with stable and ruptured carotid atherosclerotic plaques. The RNA analysis will be conducted with the microarrays.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Patients undergoing carotid endarterectomy or stenting (endovascular) for established clinical criteria
* Age > 18 years
* Male or Female
* English speaking
* Patients must sign written informed consent form

Inclusion Criteria (Controls):

* A spouse or sibling of a Patient Subject
* Age > 18 years
* Male or Female
* English speaking
* Control-Subject must sign a written informed consent form

Exclusion Criteria (Patients):

* Previous history of carotid artery surgery (endovascular or open) on the same side
* Previous cervical radiation
* Patients not felt be suitable for carotid endarterectomy or stenting (endovascular)
* Patients with impaired consent capacity
* Contraindication to MRI scans (impaired renal function, need for sedative medication during scans, inability to lie in scanner for 60 minutes)
* Prisoner status

Exclusion Criteria (Controls):

* Control-Subjects with impaired consent capacity
* Prisoner status
* Previous history of Stroke or TIAs
* Previous history of carotid artery surgery (endovascular or open)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the population of patients scheduled to undergo carotid endarterectomy or stenting for established clinical indications. These indications include patients scheduled to have a carotid endarterectomy or stenting due to the presence of a high-grade atherosclerotic cervical internal carotid artery stenosis with or without clinical symptoms, following the ACAS or NASCET criteria (carotid artery stenosis of 60% or greater without clinical symptoms; stenosis 70% or greater with clinical symptoms).
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Ultrasound Strain Measurements (Gray Scale Median Value) on Carotid Plaques | baseline (pre-surgery), 1 year follow up
  Ultrasound Radio frequency (RF) data will be acquired on patients, using both one-dimensional (1D) and two-dimensional (2D) wobbler and/or matrix array transducers to obtain four-dimensional (3D + time) RF data sets. The hypothesis is that plaques which have a lower gray scale median value and which during deformations of the cardiac cycles show larger stress concentrations in these regions are more vulnerable to rupture.
Change in In-vivo velocity measured by Transcranial Doppler (TCD) | baseline (pre-surgery), 1 year follow up
  TCD will be utilized to acquire in-vivo velocity (peak systolic, mean, and end diastolic velocity information) measurements of blood flow in the right and left middle cerebral arteries.
Change in Systolic to diastolic ratio measured by transcranial Doppler (TCD) | baseline (pre-surgery), 1 year follow up
  TCD will be utilized to acquire systolic to diastolic (S/D) ratio of blood flow in the right and left middle cerebral arteries.
Change in Pulsatility index measured by transcranial Doppler (TCD) | baseline (pre-surgery), 1 year follow up
  TCD will be utilized to acquire pulsatility index (PI) measurements of blood flow in the right and left middle cerebral arteries.
Change in Resistive index measured by transcranial Doppler (TCD) | baseline (pre-surgery), 1 year follow up
  TCD will be utilized to acquire resistive index (RI) measurements of blood flow in the right and left middle cerebral arteries.
Histopathologic classification of carotid atherosclerotic plaque after removal for plaque ulceration | obtained day of surgery
  Histologic classification of plaques is made using the updated classification of atherosclerotic plaques recommended by the American Heart association.
Change in Impairment Index - General Cognitive Morbidity | baseline (pre-surgery), 1 year follow up
  General cognitive morbidity will be derived by comparison of the Kaufman 4-subtest IQ and NART. The NART is brief standardized test that assesses an individual's ability to read irregular words (e.g., subtle). Performance on this test has been shown to be highly correlated with years of formal education and premorbid intellectual ability as assessed by traditional intelligence tests. Performance on NART will serve as a comparison against which to compare current IQ as determined by a brief 4-subtest version of the WAIS-R. This abbreviated IQ measure has been demonstrated to have very high correlation (r > .95) with the complete standard WAIS-R Full Scale IQ. Comparison of predicted versus obtained IQ will provide a measure of potential cognitive decline to be used in comparison of groups at study entry.

SECONDARY OUTCOMES:
Change in Impairment Index - Number of Abnormal Test Scores | baseline (pre-surgery), 1 year follow up
  The 60-minute cognitive screen is the most thorough assessment with the greatest sensitivity to detect the cognitive disruption associated with vascular cognitive impairment (VCI). The cognitive domains to be assessed include executive function and activation, visuospatial ability, language/lexical retrieval, and memory/learning, for a total of 10 tests. A summary impairment index will be derived for each participant and include the proportion of abnormal test scores.
Change in Impairment Index - Cognitive Domain Z-scores | baseline (pre-surgery), 1 year follow up
  A summary impairment index will be derived for each participant in part using composite cognitive domain z-scores (executive function, visuospatial, language, memory).

OTHER OUTCOMES:
Thickness of the fibrous cap | obtained day of surgery
  Examination of fibrous cap of the atherosclerotic plaque to measure thickness.
Number of vascular channels | obtained day of surgery
  Histopathologic examination of vascular channels to determine the number of channels in the fibrous cap vs the plaque proper.
Percent diameter stenosis measured with MRI | baseline (pre-surgery)
  The percent diameter stenosis will be determined with NASCET criteria.
Maximum Plaque Thickness measured with MRI | baseline (pre-surgery)
  Maximum plaque thickness was measured in the transverse plane, perpendicular to the center axis of the lumen
Number of ulcerations measured with MRI | baseline (pre-surgery)
  Ulceration will be determined by using a size threshold of 1 mm
Intraluminal Thrombus measured with MRI | baseline (pre-surgery)
  Intraluminal thrombus will be determined by a central filling defect
Thinnest area of the enhancing FC | baseline (pre-surgery)
  The thinnest area of the enhancing FC will be recorded with FC fissuring being defined as full thickness defects
Carotid intraplaque hemorrhage (IPH) | baseline (pre-surgery)
  Carotid IPH will be defined by MPnRAGE-positive plaque with ≥2-fold signal compared with the sternocleidomastoid muscle
Volumetrics | baseline (pre-surgery)
  Total volumes of plaque, lipid-rich necrotic core (LRNC), IPH, and neovascularity will be determined quantitatively with volumes manually segmented from multi-contrast scans
White Matter Hyperintensity (WMH) Volumes | baseline (pre-surgery)
  From brain MRI scans, WMH volume will be evaluated using semi-automated segmentation of T2-FLAIR images.
Hemoglobin A1C | baseline
High-sensitivity C-reactive protein (hs-CRP) | baseline
Fasting Lipid Panel | baseline
Compare DNA between blood, plaque, and genes | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Dempsey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Jackson DC, Mitchell CC, Varghese T, Hermann BP, Kliewer MA, Dempsey RJ. Estimation of ultrasound strain indices in carotid plaque and correlation to cognitive dysfunction. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:5627-30. doi: 10.1109/EMBC.2014.6944903. PMID 25571271
- [Background] Wang X, Jackson DC, Varghese T, Mitchell CC, Hermann BP, Kliewer MA, Dempsey RJ. Correlation of cognitive function with ultrasound strain indices in carotid plaque. Ultrasound Med Biol. 2014 Jan;40(1):78-89. doi: 10.1016/j.ultrasmedbio.2013.08.001. Epub 2013 Oct 11. PMID 24120415
- [Background] Wesley UV, Vemuganti R, Ayvaci ER, Dempsey RJ. Galectin-3 enhances angiogenic and migratory potential of microglial cells via modulation of integrin linked kinase signaling. Brain Res. 2013 Feb 16;1496:1-9. doi: 10.1016/j.brainres.2012.12.008. Epub 2012 Dec 14. PMID 23246924
- [Background] McCormick M, Varghese T, Wang X, Mitchell C, Kliewer MA, Dempsey RJ. Methods for robust in vivo strain estimation in the carotid artery. Phys Med Biol. 2012 Nov 21;57(22):7329-53. doi: 10.1088/0031-9155/57/22/7329. Epub 2012 Oct 18. PMID 23079725
- [Background] Rocque BG, Jackson D, Varghese T, Hermann B, McCormick M, Kliewer M, Mitchell C, Dempsey RJ. Impaired cognitive function in patients with atherosclerotic carotid stenosis and correlation with ultrasound strain measurements. J Neurol Sci. 2012 Nov 15;322(1-2):20-4. doi: 10.1016/j.jns.2012.05.020. Epub 2012 Jun 1. PMID 22658531
- [Background] Dempsey RJ, Vemuganti R, Varghese T, Hermann BP. A review of carotid atherosclerosis and vascular cognitive decline: a new understanding of the keys to symptomology. Neurosurgery. 2010 Aug;67(2):484-93; discussion 493-4. doi: 10.1227/01.NEU.0000371730.11404.36. PMID 20644437
- [Background] Shi H, Varghese T, Mitchell CC, McCormick M, Dempsey RJ, Kliewer MA. In vivo attenuation and equivalent scatterer size parameters for atherosclerotic carotid plaque: preliminary results. Ultrasonics. 2009 Dec;49(8):779-85. doi: 10.1016/j.ultras.2009.06.004. Epub 2009 Jul 3. PMID 19640556
- [Background] Shi H, Varghese T, Dempsey RJ, Salamat MS, Zagzebski JA. Relationship between ultrasonic attenuation, size and axial strain parameters for ex vivo atherosclerotic carotid plaque. Ultrasound Med Biol. 2008 Oct;34(10):1666-77. doi: 10.1016/j.ultrasmedbio.2008.02.014. Epub 2008 May 19. PMID 18490099
- [Background] Shi H, Tu H, Dempsey RJ, Varghese T. Ultrasonic attenuation estimation in small plaque samples using a power difference method. Ultrason Imaging. 2007 Jan;29(1):15-30. doi: 10.1177/016173460702900102. PMID 17491296
- [Background] Tureyen K, Vemuganti R, Salamat MS, Dempsey RJ. Increased angiogenesis and angiogenic gene expression in carotid artery plaques from symptomatic stroke patients. Neurosurgery. 2006 May;58(5):971-7; discussion 971-7. doi: 10.1227/01.NEU.0000210246.61817.FE. PMID 16639334
- [Background] Vemuganti R, Dempsey RJ. Increased expression of genes that control ionic homeostasis, second messenger signaling and metabolism in the carotid plaques from patients with symptomatic stroke. J Neurochem. 2006 Apr;97 Suppl 1:92-6. doi: 10.1111/j.1471-4159.2005.03516.x. PMID 16635256
- [Background] Vemuganti R, Dempsey RJ. Carotid atherosclerotic plaques from symptomatic stroke patients share the molecular fingerprints to develop in a neoplastic fashion: a microarray analysis study. Neuroscience. 2005;131(2):359-74. doi: 10.1016/j.neuroscience.2004.08.058. PMID 15708479
- [Background] Shi H, Mitchell CC, McCormick M, Kliewer MA, Dempsey RJ, Varghese T. Preliminary in vivo atherosclerotic carotid plaque characterization using the accumulated axial strain and relative lateral shift strain indices. Phys Med Biol. 2008 Nov 21;53(22):6377-94. doi: 10.1088/0031-9155/53/22/008. Epub 2008 Oct 21. PMID 18941278
- [Derived] Dempsey RJ, Varghese T, Jackson DC, Wang X, Meshram NH, Mitchell CC, Hermann BP, Johnson SC, Berman SE, Wilbrand SM. Carotid atherosclerotic plaque instability and cognition determined by ultrasound-measured plaque strain in asymptomatic patients with significant stenosis. J Neurosurg. 2018 Jan;128(1):111-119. doi: 10.3171/2016.10.JNS161299. Epub 2017 Mar 10. PMID 28298048
- [Derived] Mitchell CC, Stein JH, Cook TD, Salamat S, Wang X, Varghese T, Jackson DC, Sandoval Garcia C, Wilbrand SM, Dempsey RJ. Histopathologic Validation of Grayscale Carotid Plaque Characteristics Related to Plaque Vulnerability. Ultrasound Med Biol. 2017 Jan;43(1):129-137. doi: 10.1016/j.ultrasmedbio.2016.08.011. Epub 2016 Oct 5. PMID 27720278